CLINICAL TRIAL: NCT05799963
Title: A Prospective Multicenter Single Arm Trial to Assess the Safety and Effectiveness of Additional Sizes of the BioMatrix AlphaTM (Cobalt Chromium Biolimus A9TM Drug-eluting Stent) - ALPHA LONG Study
Brief Title: ALPHA LONG Study- BioMatrix AlphaTM Stent Study in Patients With CAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biosensors Europe SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-EU-03
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, open-label single-arm study. Prospective, multi-center, open-label single-arm study designed to enroll 85 patients in up to 15 centers in up to 3 European countries.
  All patients will be followed up for 9 months. The "BMX Alpha Registry" study will serve as reference and historic comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BioMatrix Alpha (Experimental): All patients will receive the BioMatrix Alpha as per treatment.
  Interventions: Device: BioMatrix Alpha

INTERVENTIONS:
Device: BioMatrix Alpha — Patient will be treated with BioMatrix Alpha

SUMMARY:
Prospective, multi-center, open-label single-arm study designed to enroll 85 patients in up to 15 centers in up to 3 European countries.

All patients will be followed up for 9 months. The "BMX Alpha Registry" study will serve as reference and historic comparator.

DETAILED DESCRIPTION:
The objective of this study is to evaluate if PCI performed using the additional sizes of the BioMatrix AlphaTM stent results in similar safety and efficacy outcomes as the currently approved (CE marked) sizes of BioMatrix Alpha.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written informed consent
2. Patient is at least 18 years old
3. Patients scheduled to undergo PCI of a de novo lesion(s) with reference vessel diameter and lesion length suitable for treatment with at least one study device
4. Patients who agree to comply with the follow up requirements
5. Patients with a life expectancy of > 1 year at time of consent
6. Patients eligible to receive for ≥6 months either dual anti-platelet therapy (DAPT, i.e. 75 mg clopidogrel or another P2Y12 inhibitor per choice of the investigator, and 75-100 mg aspirin) or a combination of an oral anti-coagulant (Vitamin K antagonist or novel anti-coagulant) and a single anti-platelet agent
7. Hemodynamically stable patients

Exclusion Criteria:

1. Inability to provide informed consent
2. Currently participating in another clinical trial
3. Planned surgery ≤6 months of PCI unless DAPT or combination anti-thrombotic/anti-platelet therapy is maintained throughout the peri-surgical period
4. Planned use of additional stents other than BioMatrix AlphaTM during the index procedure.
5. Patients with a life expectancy of < 1 year
6. Known hypersensitivity or contraindication to aspirin, clopidogrel (or to any other P2Y12 inhibitor if applicable), cobalt chromium, zinc, Biolimus A9 or a sensitivity to contrast media, which cannot be adequately pre-medicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Target Lesion Failure (TLF) | at 9 months after index procedure
  Primary endpoint is the rate of Target Lesion Failure (TLF) at 9 months defined as cardiovascular death or target vessel myocardial infarction or clinically indicated target lesion revascularization (TLR)

SECONDARY OUTCOMES:
Number of participants with Cardiovascular Death (CD) | at 9 months after index procedure
  Incidence
Number of participants with Target Vessel Myocardial Infarction | at 9 months after index procedure
  Target Vessel Myocardial Infarction (TV-MI)
Number of participants with Clinically indicated Target Lesion Revascularization | at 9 months after index procedure
  Clinically indicated Target Lesion Revascularization (ci-TLR)
Number of participants with Target Vessel Revascularization | at 9 months after index procedure
  Target Vessel Revascularization (TVR)
Number of participants with Stent thrombosis (definite and/or probable) | at 9 months after index procedure
  incidence
Number of of participants with All-cause mortality | at 9 months after index procedure
  incidence

CONTACTS AND LOCATIONS:
Overall Officials: Scot Garg, Professor, Principal Investigator — Royal Blackburn Hospital, Haslingden Rd, Blackburn BB2 3HH, UK
Locations (9):
- Germany (3):
  - Klinikum Bielefeld, Bielefeld
  - Krankenhaus Buchholz, Buchholz
  - Klinikum Lippe GmbH, Detmold
- United Kingdom (6):
  - University Hospitals Birmingham (UHB), Birmingham
  - Royal Blackburn Hospital, Blackburn
  - Hull University Teaching Hospitals (HUTH), Hull
  - United Lincolnshire Hospitals (ULH), Lincoln
  - The Grange University Hospital, Newport, Newport
  - Royal Albert Edward Infirmary, Wigan

IPD SHARING:
Plan to Share IPD: No